CLINICAL TRIAL: NCT02931721
Title: Treatment of Severe Male Infertility - Predictive Factors (Imaging)
Acronym: TESE-MRI
Status: Completed | Type: Observational
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Rauni Klami, MD, Turku University Hospital
Other Study IDs: TESE-MRI
Record Dates: First submitted 2016-10-05; First posted 2016-10-13 (Estimated); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Male Infertility
Keywords: Azospermia; Micro Dissection Testicular Sperm Extraction; Male infertility; Testis; MRI
MeSH Terms: conditions — Infertility, Male; Azoospermia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- MRI Positive: Men with sperm found in MD-TESE
  Interventions: Diagnostic Test: MRI
- MRI Negative: Men with no sperm found in MD-TESE
  Interventions: Diagnostic Test: MRI
- Control group: No intervention, fertile
  Interventions: Diagnostic Test: MRI

INTERVENTIONS:
Diagnostic Test: MRI — Pelvis MRI

SUMMARY:
Testes of men with non-obstructive azoospermia (NOA) are imaged using MRI to find potential differences depending on the outcome, ie. sperm recovery in consequent microdissection testicular sperm extraction (MD-TESE).

DETAILED DESCRIPTION:
Sperm recovery rate in non-obstructive azoospermia (NOA) men is 43% in Turku University Hospital, depending on the diagnosis leading to NOA. To date, there are no known parameters known to differentiate between successful and unsuccessful sperm recovery.

MRI is performed on men prior to the operation, and the objective is to compare the functional parameters assessed by magnetic resonance imaging between the group of men with positive and the men with negative sperm recovery in testicular microdissection sperm extraction (MD-TESE).

ELIGIBILITY:
Inclusion Criteria:

* non obstructive azospermia

Exclusion Criteria:

* malignancy
* contraindication for fertility treatment

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Azoospermic men scheduled for MD-TESE
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2023-07 (Actual); Study Completion 2023-07 (Actual)

PRIMARY OUTCOMES:
Functional difference in testicular MRI depending on MD-TESE outcome (=sperm recovery) | Baseline/ pre-invention
  ADC differences by diagnosis and outcome

CONTACTS AND LOCATIONS:
Overall Officials: Antti Perheentupa, MD,PhD, Study Director — Turku University Hospital
Locations (2):
- Finland (2):
  - Turku University Hospital, Dept of Obst and Gyn, Turku
  - Dept of Obst and Gyn, Turku

IPD SHARING:
Plan to Share IPD: No